CLINICAL TRIAL: NCT06853912
Title: A Phase 2 Single-site, Double-blind, Placebo-controlled, Randomized Clinical Trial With an Open-label Extension Phase to Examine the Safety, Subjective Experiences, Acute Effects, and Suitability of Psilocybin Combined With Psychological Support (Psi-PS) for Military Veterans and First Responders With Co-occurring Alcohol Use Disorder (AUD) and Posttraumatic Stress Disorder (PTSD)
Brief Title: Psilocybin With Psychological Support (Psi-PS) for Military Veterans and First Responders With Co-occurring PTSD & Alcohol Use Disorder (AUD)
Acronym: Psi-PS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Brashares Sackett (Other)
Collaborators: Washington State Legislation (Unknown)
Responsible Party: Sponsor-Investigator, Nathan Brashares Sackett, Addiction Psychiatrist, Assistant Professor, University of Washington
Organization: University of Washington (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00021194
Record Dates: First submitted 2024-12-11; First posted 2025-03-03 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder (AUD); PTSD
Keywords: Psilocybin; Psychological Support; PTSD; AUD; Military Veterans and First Responders; Psychedelics; Vet; Veteran; Post-Traumatic Stress Disorder; Alcohol; Alcohol Use Disorder; Post Traumatic Stress Disorder; Military; Military Veterans; First Responders; Healthcare Workers
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Psilocybin; maltodextrin

STUDY DESIGN:
Intervention Model Description: A single-site, double-blinded, placebo-controlled, randomized clinical trial with an open-label extension phase assessing safety in two conditions: (1) 25 mg of psilocybin combined with nondirective psychological support (Psi-PS); and (2) placebo and nondirective psychological support.
Who Masked: Participant, Investigator
Masking Description: The study team and participants will remain masked until 1-month post-Drug Administration Session follow-up data are collected from each participant. At the end of this visit, all parties will be unmasked and those revealed to have received placebo will be invited to participate in an open-label extension where they repeat two preparation sessions, the drug administration session, and three integration sessions (Visits 4-9) with psilocybin before moving into long-term follow-up at 12- and 24-weeks post-Drug Administration Session. If a participant in the placebo arm declines to participate in the Open-Label Extension, they will move into the 12- and 24-week post-Drug Administration Session follow-up visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin + Nondirective Psychological Support (Experimental): The intervention is composed of two 60-minute telehealth preparation sessions (Prep 1 and Prep 2) with two facilitators; one 6-8-hour drug administration session (25 mg of oral psilocybin) in a clinical setting with the same two facilitators present; and three 60-minute telehealth integration sessions (Integration 1-3) with the same two facilitators. Ideally the entire intervention will be delivered over 6 weeks allowing for some flexibility based on schedules and logistics.
  Interventions: Drug: Psilocybin 25 mg
- Placebo + Nondirective Psychological Support (Placebo Comparator): The arm is composed of two 60-minute telehealth preparation sessions (Prep 1 and Prep 2) with two facilitators; inert placebo (25 mg of Maltodextrin) administered in a clinical setting with the same two facilitators present; and three 60-minute telehealth integration sessions (Integration 1-3) with the same two facilitators. Ideally the entire intervention will be delivered over 6 weeks allowing for some flexibility based on schedules and logistics.
  Interventions: Drug: Maltodextrin (Placebo)

INTERVENTIONS:
Drug: Psilocybin 25 mg — Botanical drug product PEX010(25) contains the drug substance, PYEX, which is primarily composed of psilocybin (delivered in a capsule)
  Other Names: PEX010; PYEX
  Arms: Psilocybin + Nondirective Psychological Support
Drug: Maltodextrin (Placebo) — 25 mg of Maltodextrin (delivered in a capsule)
  Arms: Placebo + Nondirective Psychological Support

SUMMARY:
This study is a phase 2 single-site, double-blind, placebo-controlled, randomized clinical trial with an open-label extension phase to examine the safety of psilocybin (25 mg) combined with psychological support (Psi-PS) for treatment of approximately 40 military veterans and first responders (ages 21-65) with co-occurring alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD). Psychological support is defined as providing safety, reassurance, active listening, and empathetic presence during the drug administration session in a nondirective manner. We hypothesize that Psi-PS may provide a safe treatment for participants. The primary objective of study is to characterize the safety of psilocybin combined with psychological support (Psi-PS) for individuals with co-occurring alcohol use disorder (AUD) and PTSD.

DETAILED DESCRIPTION:
There is growing evidence suggesting that psychedelic drugs, when paired with therapy, may constitute a safe and effective form of treating a diverse range of psychopathological issues such as alcohol use disorder (AUD) and PTSD (Bogenschutz et al., 2015, 2022; Dakwar et al., 2020; Grabski et al., 2022; Mitchell et al., 2021, 2023). However, to date, no studies have explored any form of psychedelic-assisted therapy in the treatment of patients with co-occurring AUD and PTSD, despite high rates of comorbidity. This study will be the first of its kind to evaluate the safety of psilocybin paired with therapy to target symptoms of comorbid AUD and PTSD. Data derived from this clinical trial will help shed light on whether Psi-PS may be safe for those suffering from both PTSD and AUD.

Taken together, we propose the following primary, secondary, and exploratory objectives:

1. Primary Objective: Characterize the safety of psilocybin combined with psychological support (Psi-PS) for participants during the drug administration session (DAS) while the drug's acute effects are ongoing, approximately 24 hours after the DAS when the drug's acute effects have subsided, and approximately one-week post-DAS.
2. Exploratory Objective: (1) Explore the subjective experiences of Psi-PS within approximately 24 hours following the DAS, i.e., when the drug's acute effects have subsided, approximately one-week following the DAS, and at follow-up at approximately three-months. (2) Assess acute effects of Psi-PS on a range of variables at baseline and weeks 1, 2, 4, 12, and 24 post-DAS; (3) Further, assess suitability at baseline and approximately 4-weeks post-DAS.

This study is a single-site, double-blinded, placebo-controlled, randomized clinical trial with an open-label extension phase assessing safety in two conditions: 1. Psi-PS (psilocybin combined with psychological support); and 2. placebo and nondirective psychological support. The study will last approximately 26-32 weeks and is composed of two preparation sessions; one Drug Administration Session (DAS), where 25 mg of oral psilocybin (PEX010) or inert placebo (PCB2) is administered in a clinical setting with two facilitators present; and three integration sessions. Placebo conditions will receive the same psychological support but will receive an inert placebo. 4-weeks after DAS, the study will be unblinded and those who received placebo will be offered Psi-PS for the open-label extension phase, following the same procedures. The intended sample size for the study is approximately 40 military veterans and first responders (ages 21-65) with co-occurring alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD). Study drug shipments will arrive on-site pre randomized by the manufacturer, and double-blinding will be maintained throughout the study by using a placebo that is designed to have similar physical characteristics as the study drug. All participants will then be followed for a total of 6 months (24 weeks) following the DAS to assess durability of potential effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 21-65 who meet criteria for current DSM-5 diagnosis of AUD and PTSD as determined by the Alcohol System Checklist and CAPS-5.
2. Are either a US military Veteran or are currently employed as a first responder, including EMT, paramedic, firefighter, or law enforcement officer.
3. Report wanting to stop or decrease drinking and are willing to abstain from alcohol for the week prior to receiving any study drug.
4. Are English-speaking.
5. Must be willing to use contraception throughout the duration of the study. This applies to anyone, regardless of biological sex, who can cause pregnancy or become pregnant themselves.
6. Have a friend or family member who can pick them up and stay with them overnight after the DAS and who agrees to share contact information with the research team.
7. Have a primary care provider.
8. Have access to stable internet and either smart phone or computer.
9. Are willing to disclose medication use, supplement use, and interventions they are currently enrolled in; and commit to all study-related activities and follow-up sessions.
10. For the drug administration session, participants must be willing to reduce alcohol intake to be alcohol-free for 24 hours before DAS, fast after midnight before DAS, avoid caffeine and nicotine 2 hours before and 6-8 hours after DAS, and avoid driving for 24 hours post-DAS.
11. Must be locally accessible to the University of Washington for multiple in-person study visits.
12. Must have a friend or someone else the participant trusts to stay with them overnight for the evening following the DAS.

Exclusion Criteria:

1. A reported history of known medical conditions that would preclude safe participation in the trial, including the following:

   * seizure disorder,
   * coronary artery disease,
   * history of arrhythmia or known valvopathy,
   * heart failure,
   * cerebrovascular accident,
   * severe asthma
   * pulmonary hypertension,
   * hyperthyroidism,
   * stenosing peptic ulcer,
   * pyloroduodenal obstruction,
   * symptomatic prostatic hypertrophy,
   * bladder-neck obstruction.
2. Clinical findings on screening, including:

   * significantly impaired liver function found in labs in prior 45-days or at screening
   * uncontrolled hypertension (above 165/95 mmHg at screening)
   * Serious ECG abnormalities measured at or within 45-days of screening (e.g., evidence of ischemia, myocardial infarction, QTc prolongation (QTc > 0.45 seconds for men, QTc > 0.47 seconds for women).
3. Reported history or findings on SCID-CT of known exclusionary psychiatric conditions, including schizophrenia, schizoaffective disorder, bipolar disorder type I or type II.
4. A reported history of a serious suicide attempt (SSA) in previous 12-months.
5. A reported history of a personality disorder at time of screening.
6. A reported family history of schizophrenia or schizoaffective disorder (first- or second-degree relatives), or bipolar disorder type 1 (first degree relatives).
7. Currently using SSRIs, SNRIs, MAOIs, TCAs, antipsychotics, lithium, stimulants, or other psychedelics.
8. Currently engaged in CBT, DBT, EMDR, psychoanalytic/psychodynamic therapy, MBSR, or unapproved group therapies, except for peer support groups.
9. Cognitive impairment (Folstein Mini Mental State Exam score < 26).
10. A reported lifetime history of hallucinogen use disorder (per DSM-5).
11. A reported history of cocaine, psychostimulant, or opioid use disorder defined by DSM-5 in the past 12 months, or currently utilizing full-agonist (methadone) or partial-agonist (buprenorphine) for OUD.
12. Current or historical abuse of psychedelic/hallucinogenic substances (e.g. LSD, mushrooms/psilocybin, mescaline/peyote, MDMA, ketamine, ayahuasca, ibogaine, DMT, etc.) endorsed by participant or suspected by the Lead Investigator's clinical judgement.
13. Reported current non-medical use of cocaine, psychostimulants, psilocybin, or opioids (past 30 days).
14. A reported history of significant alcohol withdrawal (CIWA-Ar score greater than 7) or a history of severe alcohol withdrawal, including delirium tremens, withdrawal seizures or any acute hospitalization related to alcohol withdrawal. Participants presenting at screening in withdrawal may be referred for detoxification and reassessed within 30 days.
15. Serious abnormalities of complete blood count (CBC) or chemistries found at or within 45-days of screening.
16. Currently enrolled in another clinical trial of any kind.
17. Active legal problems with the potential to result in incarceration.
18. Pregnancy or lactation; or intention to become pregnant or cause pregnancy
19. Need to take medication with significant potential to interact with study medications (e.g., antidepressants, antipsychotics, psychostimulants, treatments for addictions, other dopaminergic or serotonergic agents, lithium, anticonvulsants) as determined by Study Physician or Lead Investigator.
20. Allergy or hypersensitivity to psilocybin.
21. High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support), or deemed not suitable for other reasons stipulated by the research team.
22. A previous diagnosis of Hallucination Perceptual Persisting Disorder (HPPD).
23. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 3 months or 5 half-lives before enrollment or is currently enrolled in the treatment stage of an investigational study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Psi-PS | Within approximately 24 hours post-DAS, i.e., when the drug's acute effects have subsided, and approximately one-week post-DAS.
  Safety of Psi-PS will be measured through the assessment of adverse events (AEs), serious adverse events (SAEs), and acute suicidality using the Columbia Suicide Severity Rating Scale (C-SSRS).

SECONDARY OUTCOMES:
Subjective Experiences | On the day of the DAS, 1-week post-DAS, and 3-months post-DAS
  Describe the subjective experiences of psilocybin combined with psychological support (Psi-PS) for individuals with alcohol use disorder (AUD) and PTSD with qualitative data analyses.

OTHER OUTCOMES:
Changes in Alcohol Use and PTSD Symptom Severity, Suitability, and Acute Effects | 1-, 3-, and 6-months post-treatment between psilocybin and placebo groups
  Compare changes in alcohol use at 1-, 3-, and 6-months post-treatment between psilocybin and placebo groups; Compare changes in PTSD symptom severity at 1-, 3-, and 6-months post-treatment between psilocybin and placebo groups; Assess the suitability of Psi-PS for individuals with AUD and PTSD; Characterize the acute effects of Psi-PS for individuals with AUD and PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan B Sackett, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Center for Novel Therapeutics in Addiction Psychiatry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No